CLINICAL TRIAL: NCT03597685
Title: ProLyPhy-GEP : Pesticide Associated Lymphomas: Expression of Treatment Resistance Genes
Brief Title: Pesticide Associated Lymphomas: Expression of Treatment Resistance Genes
Acronym: ProLyPhy-GEP
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0010
Record Dates: First submitted 2018-01-16; First posted 2018-07-24 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-03

CONDITIONS: Lymphoma Diffuse Large B-cell
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lymphomagenesis is partially known, and some risk factor are identified like those inducing immune deficiencies: chronic exposure to HIV, immune suppressor therapies or commun variable immunodeficiency. Parts of the mechanisms leading to NHL development after pesticide exposure are the disruption of immune surveillance against cancer cell. Pro-oncogenic action of metabolites is the most important mechanisms of action for pesticides. Thus, pesticides are metabolized in pro-oxidant compounds disturbing the redox homeostasis in the haematopoietic and immune cells precursors, promoting proliferation and survival, and inducing DNA breaks. Some of them induce direct DNA breaks and non-conform reparation, leading to activation of oncogenes; and other induces transcription factors for oncogenic signalling pathways. DNA reparation and adaptation to a higher ROS level are associated with resistance against cytotoxic chemotherapy treatment with induction of detoxification mechanism by tumour cells.

That DNA repair pathways, which are targeted by chemotherapy could also explain a part of chemo-resistance. It was therefore suggested that DLBCL dependence to specific DNA repair pathways could be targeted to hamper repair of intrinsic DNA damage occurring during B-lymphoma cells proliferation or to increase DNA damage induced by chemotherapy.

DETAILED DESCRIPTION:
Occupational exposure to pesticides is associated with higher incidence of non-Hodgkin lymphoma (NHL), including diffuse large B-cell lymphoma (DLBCL) The relative risk for NHL after occupational exposure to pesticide is 1.5 to 3, with little variation according to NHL subtypes. DLBCL is one of the most frequent subtypes of NHL and characterized by aggressive presentation. DLBCL is treated by chemotherapy based on anthracyclines combined with an anti-CD20 monoclonal antibody allowing complete response and long term remission in 65-70% of patients. The response rate to treatment and clinical outcome is depending of the DLBCL subtype. There are 3 of them depending of the cell of origin (germinal centre B cell or activated B cell), and the anatomical location (primary mediastinal) identified by molecular gene expression profile. The activated B cell subtype have a worse outcome.

Lymphomagenesis is partially known, and some risk factor are identified like those inducing immune deficiencies: chronic exposure to HIV, immune suppressor therapies or commun variable immunodeficiency. Parts of the mechanisms leading to NHL development after pesticide exposure are the disruption of immune surveillance against cancer cell. Pro-oncogenic action of metabolites is the most important mechanisms of action for pesticides. Thus, pesticides are metabolized in pro-oxidant compounds disturbing the redox homeostasis in the haematopoietic and immune cells precursors, promoting proliferation and survival, and inducing DNA breaks. Some of them induce direct DNA breaks and non-conform reparation, leading to activation of oncogenes; and other induces transcription factors for oncogenic signalling pathways. DNA reparation and adaptation to a higher ROS level are associated with resistance against cytotoxic chemotherapy treatment with induction of detoxification mechanism by tumour cells.

That DNA repair pathways, which are targeted by chemotherapy could also explain a part of chemo-resistance. It was therefore suggested that DLBCL dependence to specific DNA repair pathways could be targeted to hamper repair of intrinsic DNA damage occurring during B-lymphoma cells proliferation or to increase DNA damage induced by chemotherapy.

The investigators hypothesize that actions of pesticides on DNA and redox homeostasis are critical events during lymphomagenesis. We supposed that specific mechanisms of DNA repair and antioxidant defences induced by pesticides exposure are implicated in the chemo-resistance in DLBCL patients.

There might be a negative impact of professional exposure to pesticide on treatment response.

In this search, the investigators will explore a comprehensive view of both lymphomagenesis and adverse prognosis of pesticide-exposed DLBCL. The investigators plan to analyse the molecular profile of B-lymphoma cells from pesticide-exposed patients, to better understand biological mechanisms underlying lymphomagenesis as well as chemotherapy resistance

ELIGIBILITY:
Inclusion Criteria:

Adults treated for diffuse large B-cell lymphoma:

* Diagnosed between 2010 and 2015
* Included in ProLyPhy search
* Having received R-CHOP immuno-chemotherapy
* Supported in health facilities in Languedoc-Rousillon

Exclusion criterion:

NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults treated for diffuse large B-cell lymphoma:
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
genes implicated in chemoresistance of diffuse large B-cell lymphoma | 1 day
  Use of excesses of the biopsy made as part of the care for the diagnostic of the lymphoma for identify genes implicated in chemoresistance of DLBCL

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain LAMURE, CCA, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC